CLINICAL TRIAL: NCT07142187
Title: The Effect of Electro-thumbtack Needle on Live Birth Rate in Patients With Ovarian Reserve Dysfunction (DOR): a Multicenter Randomized Controlled Clinical Trial
Brief Title: The Clinical Trial of Electro-thumbtack Needle on Live Birth Rate in Patients With Ovarian Reserve Dysfunction (DOR)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Dongmei Huang, Clinical Professor of Integrated Traditional Chinese and Western Medicine at Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJ-IRB202508011
Record Dates: First submitted 2025-04-06; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Diminished Ovarian Reserve (DOR)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electro-thumbtack needle group (Experimental): Electro-thumbtack needle is a sterile needle with a special conductive chip that can conduct electricity. Electro-thumbtack needle enhances the stimulation effect on acupoints by introducing pulsed microcurrents, and is a long-lasting needle retention therapy with stronger stimulation effect than ordinary acupressure.
  Interventions: Other: electro-thumbtack needle
- Placebo group (Placebo Comparator): Placebo electro-thumbtack needle use insulated soft silk threads instead of needle bodies, making their appearance, shape, and color no different from real electro-thumbtack needle, but without needle like effects; Placebo electro-thumbtack needle also do not have the conductivity of true electric needles (silk threads are insulated); The placebo conductive patch used in the control group, although having the same appearance as the treatment group, is a specially insulated control substance. Therefore, even if the pulse generator is turned on and adjusted to medium intensity, the patient still receives zero current stimulation intensity.
  Interventions: Other: placebo electro-thumbtack needle

INTERVENTIONS:
Other: electro-thumbtack needle — The treatment acupoints include bilateral ovarian acupoints, Guan Yuan (CV4), bilateral Shen Shu (BL23), bilateral waist and eye acupoints (EX-B7), bilateral San Yin Jiao (SP6), and bilateral Zu San Li (ST36), totaling 11 acupoints. Among them, the bilateral ovarian acupoints and bilateral waist eye acupoints (EX-B7) were treated with electro-thumbtack needle. Other acupoints were treated with thumbtack needle.Choose a sparse and dense waveform, adjust the intensity to the maximum patient can tolerate, and stimulate for 30 minutes each time. After the stimulation is completed, remove the electrode patch and electroacupuncture device, and keep the electric needle at the acupoint for another 3 days.During the needle retention period, the electric needles at the bilateral ovarian acupoints and bilateral waist and eye acupoints were alternately stimulated once every other day using an electroacupuncture device for 30 minutes each time.
  Arms: electro-thumbtack needle group
Other: placebo electro-thumbtack needle — The control group selected acupoints that were the same as the treatment group. Bilateral ovarian acupoints and bilateral waist and eye acupoints are treated with placebo electro-thumbtack needle, while other acupoints are treated with placebo electro-thumbtack needle. The treatment methods for placebo electro-thumbtack needle and placebo thumbtack needle are the same as those for the treatment group.
  Arms: Placebo group

SUMMARY:
This study will include 246 patients with ovarian reserve dysfunction (DOR), who will be randomly divided into a treatment group and a control group, with 123 patients in each group. The treatment group will receive electro-thumbtack needle treatment, while the control group will receive placebo electro-thumbtack needle treatment. Both groups will receive a treatment course of 3 menstrual cycles. This study evaluates the effect of electrocautery on the live birth rate of patients with DOR.

ELIGIBILITY:
Inclusion Criteria:

* The age range is 18-40 years old;
* Meets the diagnostic criteria for DOR as follows: ① AMH<1.1 ng/ml; ② 10 U/L < FSH < 25U/L or FSH/LH > 3.6; ③ The total number of follicles (AFC) in both basal sinuses is less than 7. If any two of the above criteria (①②③) are met, it can be diagnosed as DOR.
* At least one side of the patient's fallopian tube is unobstructed;
* The semen routine examination of the patient's spouse is normal;
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Chromosomal or genetic abnormalities in either the female or male partner;
* Women with blocked fallopian tubes on both sides;
* Have a history of ovarian surgery, such as ovarian teratoma or ovarian chocolate cyst surgery;
* The female party suffers from uncorrected endocrine disorders such as simple hyperthyroidism or hypothyroidism, hyperprolactinemia, and pancreatic islet dysfunction;
* Hormone resistance, diabetes, adrenal diseases, etc;
* The woman has a clearly diagnosed autoimmune disease such as systemic lupus erythematosus, rheumatoid arthritis;
* Antiphospholipid syndrome, Sjogren's syndrome, Hashimoto's thyroiditis, etc;
* The female or male partner has a history of malignant tumors and has received treatment with radiotherapy and chemotherapy;
* The woman has received acupuncture and moxibustion or press acupuncture treatment in recent 3 months;
* Those who take traditional Chinese medicine decoctions or granules during treatment;
* Men with abnormal semen examination;
* Clear diagnosis of moderate or severe adenomyosis;
* Clearly diagnose uterine fibroids with a diameter greater than 5cm;
* I do not agree to sign the informed consent form for this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 368 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 3 months
  The live birth rate is defined as the proportion of live births after 28 weeks of pregnancy, usually calculated by dividing the number of live birth cycles by the total number of patients and multiplying by 100%. This indicator is commonly used to evaluate the effectiveness of reproductive health centers or specific treatment methods, reflecting the ultimate outcome of successful pregnancy.

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 3 months
  Biochemical pregnancy, also known as subclinical miscarriage or occult miscarriage, refers to the phenomenon where the embryo fails to successfully implant on the uterine wall in the early stages, leading to termination of pregnancy.The biochemical pregnancy rate is calculated by dividing the number of biochemical pregnancies by the total number of patients.
clinical pregnancy rate | 3 months
  Clinical pregnancy refers to the presence of a gestational sac in the uterine cavity, as well as the appearance of fetal buds and primitive heartbeats, observed through ultrasound examination in the early stages of pregnancy. These signs indicate normal implantation and development of the embryo, confirming a normal intrauterine pregnancy.The clinical pregnancy rate is calculated by dividing the number of pregnancies by the total number of patients.
Threatened miscarriage rate | 3 months
  Threatened miscarriage refers to symptoms such as vaginal bleeding and abdominal pain that occur before 28 weeks of pregnancy, but at this time the cervix is not open, the membranes are intact, there is no discharge of pregnancy material, and the size of the uterus matches the gestational age. The threatened miscarriage rate is calculated by dividing the number of threatened miscarriages by the total number of patients.
abortion rate | 3 months
  The miscarriage rate is calculated by dividing the number of miscarriages by the total number of patients.
Anti Mullerian hormone (AMH) | 3 months
  Anti Mullerian hormone (AMH) is a glycoprotein hormone secreted by follicular granulosa cells in the ovary. It is of great significance in evaluating women's ovarian reserve function and can be used to assess the number and quality of follicles in the ovaries. The concentration of AMH in serum will be measured.
Antral Follicle Count (AFC) | 3 months
  Antral Follicle Count (AFC) refers to the count of antral follicles present in the ovary using ultrasound technology. Sinus follicles are small follicles with a diameter of approximately 2-9mm located in the ovary. These follicles are in the early developmental stage of the cycle and have a good correlation with women's ovarian reserve function
follicle stimulating hormone（FSH） | 3 months
  The concentration of follicle stimulating hormone（FSH） in serum will be measured. The changes in FSH levels can reflect ovarian function and ovulation status, and are of great significance for the diagnosis and monitoring of various gynecological diseases.FSH was measured on the second day of menstruation.
Luteinizing hormone (LH) | 3 months
  The concentration of Luteinizing hormone (LH) in serum will be measured. LH is a glycoprotein hormone secreted by pituitary cells, mainly acting on mature oocytes, which can induce ovulation and produce corpus luteum.LH is measured on the second day of menstruation.
estradiol（E2） | 3 months
  The concentration of estradiol（E2） in serum will be measured.The level of estradiol is commonly used to assess the reproductive health status of women, which is measured on the second day of menstruation.
Progesterone（P） | 3 months
  The concentration of Progesterone（P） in serum will be measured.Progesterone is an important progesterone mainly secreted by the corpus luteum of the ovary and also present in the adrenal cortex and placenta. Progesterone plays a crucial role in the female reproductive system, including maintaining normal menstrual cycles, promoting endometrial development, providing a suitable implantation environment for fertilized eggs, and maintaining pregnancy.
Prolactin（PRL） | 3 months
  The concentration of Prolactin（PRL） in serum will be measured.Prolactin also affects female reproductive function, such as follicle development and ovulation process
Testosterone（T） | 3 months
  The concentration of Testosterone（T） in serum will be measured.Testosterone is a steroid hormone mainly secreted by the testicles of males and ovaries of females
ZungSelf-RatingAnxietyScale（Zung-SAS） | 3 months
  Zung SAS is mainly used to evaluate an individual's anxiety symptoms and their severity.The total score range of this scale is 20 to 80 points. After conversion, the score can be used as an indicator of anxiety level - usually multiplying the original score by 1.25 and converting it into a norm score. The higher the norm score, the more severe the individual's anxiety level.
Zung Self-rating depression scale(Zung-SDS) | 3 months
  Zung SDS is mainly used to evaluate the severity and changes of individual depressive symptoms.Composed of 20 questions, the scores of each of the 20 items are added together to obtain a rough score. The standard score is equal to the integer part obtained by multiplying the coarse score by 1.25. The normal upper limit of the total gross score is 41 points, and the standard total score is 53 points.
Short form-36（SF-36） | 3 months
  SF-36， The Medical Outcomes Study - Short Form, also known as the Health Survey Short Form, is a universal measurement scale developed from the Boston Health Study in the United States. This scale consists of 36 items and is evaluated.The score range of SF-36 scale is 0-100 points, where 100 points represents the best health status and 0 points represents the worst health status.
Chinese Quality of Life Scale (CHQOL) | 3 months
  The Chinese Quality of Life Scale (CHQOL) is a new universal scale developed based on the concept of traditional Chinese medicine health, which is used for evaluation.Full score of 60, the higher the score, the higher the quality of life.
Self Rating Sleep Scale (SRSS) | 3 months
  SRSS is a tool used to screen and evaluate individual sleep problems. It consists of 10 items, each rated on a 5-point scale, with higher scores indicating more severe sleep problems. The scoring criteria for the SRSS are as follows: 10 items are rated on a scale of 1-5, with a total score range of 10-50 points. The higher the score, the more severe the sleep problem.
The Sleep Disorders Rating Scale (SDRS) | 3 months
  The Sleep Disorders Rating Scale (SDRS) is a tool used to assess an individual's sleep status over the past week.Each item has a maximum score of 3 points, and the total score can reach up to 21 points. The higher the score, the more severe the sleep disorder.
Pittsburgh Sleep Quality Index (PSQI) | 3 months
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-assessment scale used to evaluate an individual's sleep quality over the past month.The total score range of the scale is 0-21 points, with higher scores indicating poorer sleep quality.
corticotropin releasing hormone (CRH) | 3 months
  The concentration of CRH in serum will be measured.Corticotropin releasing hormone (CRH) is a forty one peptide hormone secreted by the hypothalamus. Its main function is to promote the synthesis and release of adrenocorticotropic hormone (ACTH) by the pituitary gland, thereby regulating the secretion of glucocorticoids by the adrenal cortex
norepinephrine | 3 month
  The concentration of norepinephrine in serum will be measured.
epinephrine | 3 months
  The concentration of epinephrine in serum will be measured.
5-hydroxytryptamine (5-HT) | 3 months
  The concentration of 5-hydroxytryptamine (5-HT) in serum will be measured.
gamma aminobutyric acid (GABA) | 3 months
  The concentration of gamma aminobutyric acid (GABA) in serum will be measured.
dopamine (DA) | 3 months
  The concentration of dopamine (DA) in serum will be measured.
beta endorphin (β - ET) | 3 months
  The concentration of beta endorphin (β - ET) in serum will be measured.